CLINICAL TRIAL: NCT01292941
Title: Clinical Study Evaluating Safety of a New Catheter for Urinary Intermittent Catheter in Healthy Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Product development project closed prematurely
Sponsor: Coloplast A/S (Industry)
Responsible Party: MD,PhD Per Bagi, Rigshospitalet institute/Dept.2112
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: CP065CC
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active comparator/Yellow catheter (Active Comparator): SpeediCath coated catheter
  Interventions: Device: Intermittent catheterisation
- NonCE marked intermittent catheter/red (Experimental)
  Interventions: Device: NonCE marked intermittent catheter/red
- NonCE marked intermittent catheter/green (Experimental)
  Interventions: Device: NonCE marked intermittent catheter/green
- NonCE marked intermittent catheter/Blue (Experimental)
  Interventions: Device: NonCE marked intermittent catheter/blue

INTERVENTIONS:
Device: Intermittent catheterisation — Speedicath, Intermittent catheterisation
  Other Names: SpeediCath
  Arms: Active comparator/Yellow catheter
Device: NonCE marked intermittent catheter/red — Paris, Intermittent catheterisation
  Other Names: Paris
  Arms: NonCE marked intermittent catheter/red
Device: NonCE marked intermittent catheter/green — Paris, Intermittent catheter
  Other Names: Paris
  Arms: NonCE marked intermittent catheter/green
Device: NonCE marked intermittent catheter/blue — Paris, Intermittent catheter
  Other Names: Paris
  Arms: NonCE marked intermittent catheter/Blue

SUMMARY:
To evaluate discomfort of a new coating and catheter material compared to SpeediCath (SC)

DETAILED DESCRIPTION:
Intermittent catheterization is the preferred method for emptying the bladder in patients with spinal cord injury and neurogenic bladder dysfunction.

Coloplast have developed a new intermittent catheters. In this investigation this new test catheter will be compared with SpeediCat by assessing discomfort and pain associated with catheterization of healthy men. The reason for choosing healthy men is that many catheter users do not have full feeling in their urethra and therefore can not assess the discomfort.

55 healthy men who are ≥ 18 years and have no signs of urinary tract infection and do not have abnormalities, disease or have had operational interventions in the urinary tract will be included. They are recruited through advertisements on the website www.forsoegsperson.dk.

ELIGIBILITY:
Inclusion Criteria:

* • ≥18 years

  * Male
  * Signed informed consent
  * Negative urine stix (erythrocytes, leucocytes and nitrite)

Exclusion Criteria:

* • Abnormalities, diseases or surgical procedures performed in the lower urinary tract

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Discomfort during catheterisation measured by VAS-scale (0-10) | 10 measurements in an 11 week period. 10 min after each catheterisation
  A subject is assesing a VAS scale after each catheterisation.

SECONDARY OUTCOMES:
Safety | During the investigation 11 Weeks per subject
  Safety is evalueted continues while the subjects are testing the devices
Discomfort during urination post catheterisation | 10 measurements in an 11 week period. 10 min after each catheterisation
  Subjects own assesment. Yes or no can be answered to discomfort during urination post catheterisation
Haematuria | 10 measurements in an 11 week period. 10 min after each catheterisation
  Urine test after each catheterisation, and measured on a urine stix
Handling during insertion, withdrawal | 10 measurements in an 11 week period. 10 min after each catheterisation
  Ease of use assessed by nurses, measured on a 5 point scale

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Gürtler, CTM, Study Director — Coloplast A/S
Locations (1):
- Rigshospitalet, Copenhagen, Denmark